CLINICAL TRIAL: NCT02648724
Title: An Open-Label, Multicenter Phase 1a/2a Trial Investigating the Safety, Tolerability and Antitumor Activity of Multiple Doses of Sym015, a Monoclonal Antibody Mixture Targeting MET, in Patients With Advanced Solid Tumor Malignancies
Brief Title: Sym015 (Anti-MET) in Patients With Advanced Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Sym015-01; 2016-003912-11 (EudraCT Number)
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Results first posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-04

CONDITIONS: Oncology; MET Gene Amplification; NSCLC; MET Gene Mutation; Non Small Cell Lung Cancer
Keywords: Advanced Solid Tumor Malignancies; MET Gene Amplification; MET Amplification; Wild-type; NSCLC; METex14del; Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Arms 1-4 comprises part 1 (dose-escalation), which is an as evaluation of 4 different dose levels (DL), 6, 12, 18, and 24 mg/kg. DL data from part 1 is presented as merged in the other sections. This is due to that there were no dose level toxicities reported during the study.
  Arms 5-7 comprises part 2 (dose-expansion).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1: 6 mg/kg (Experimental): Sym015 was tested in four dose titration cohorts. Patients in this cohort received 6 mg/kg. A substitute or an additional dose level could potentially be evaluated.
  Interventions: Drug: Sym015
- Part 1: 12 mg/kg (Experimental): Sym015 was tested in four dose titration cohorts. Patients in this cohort received 12 mg/kg. A substitute or an additional dose level could potentially be evaluated.
  Interventions: Drug: Sym015
- Part 1: 18 mg/kg (Experimental): Sym015 was tested in four dose titration cohorts. Patients in this cohort received 18 mg/kg. A substitute or an additional dose level could potentially be evaluated.
  Interventions: Drug: Sym015
- Part 1: 24 mg/kg (Experimental): Sym015 was tested in four dose titration cohorts. Patients in this cohort received 24 mg/kg. A substitute or an additional dose level could potentially be evaluated.
  Interventions: Drug: Sym015
- Part 2: Basket Cohort (Experimental): Patients with KRAS WT advanced solid tumor malignancies with MET-amplification were to receive Sym015 at the RP2D. Included in this group was a subset of patients who have received prior therapy with a MET-targeting TKI.
  Interventions: Drug: Sym015
- Part 2: NSCLC MET-Amplified Cohort (Experimental): Patients with advanced NSCLC with MET-amplification were to receive Sym015 at the RP2D. Patients may have received prior therapy with MET-targeting and/or EGFR-targeting agents.
  Interventions: Drug: Sym015
- Part 2: NSCLC METex14del Cohort (Experimental): Patients with advanced NSCLC with METex14del were to receive Sym015 at the RP2D. Tumors need not be MET-amplified, and patients may have received prior therapy with MET-targeting and/or EGFR-targeting agents. mutation.
  Interventions: Drug: Sym015

INTERVENTIONS:
Drug: Sym015 — Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
  Other Names: Anti-MET

SUMMARY:
This is the first study to test Sym015 in humans. The primary purpose of this study is to see if Sym015 is safe and effective for patients with advanced solid tumor malignancies without available therapeutic options.

DETAILED DESCRIPTION:
In the first part of the study (Part 1, dose-escalation), Sym015 was evaluated for safety and tolerability. Additionally, the recommended Phase 2 dose (RP2D) was to be determined. Sym015 was given at different dose levels on an every second week (Q2W) dosing schedule. Each patient was given one single weight based dose level.

In the second part of the study (Part 2, dose-expansion), dosing was to be at the RP2D on a Q2W dosing schedule. Three cohorts were included:

* Basket Cohort: Patients with KRAS wild-type (WT) advanced solid tumor malignancies with MET-amplification and without therapeutic options. Patients must have no prior therapy with MET-targeting agents, except a subset of patients having received prior therapy with a MET-targeting tyrosine kinase inhibitor (TKI). As of December 2018, accrual to this cohort was suspended.
* Non-Small Cell Lung Carcinoma (NSCLC) MET-Amplified Cohort: Patients with advanced NSCLC with MET-amplification, and without available therapeutic options. Patients may have received prior therapy with MET-targeting and/or epidermal growth factor receptor (EGFR)-targeting agents.
* NSCLC with MET exon 14 skipping alteration (METex14del) Cohort: Patients with advanced NSCLC METex14del, and without therapeutic options. Tumors need not be MET-amplified, and patients may have received prior therapy with MET-targeting and/or EGFR-targeting agents.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Life expectancy >3 months assessed during Screening.
* Documented (histologically- or cytologically-proven) solid tumor malignancy that is locally advanced or metastatic, and that is refractory to standard therapy or for which no standard therapy is available or accessible.
* If female and of childbearing potential: a negative pregnancy test.
* Male or female: either not of childbearing potential or agreeing to use a medically effective method of contraception as per institutional standards during the trial and for 4 months after the last dose of trial drug.
* Part 1 ONLY: Tumor documented to be KRAS WT by local assessment.
* Part 2 ONLY:

  * Measurable disease according to RECIST v1.1 that has been confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) within 4 weeks prior to Cycle 1/Day 1 (C1/D1).
  * Basket Cohort ONLY:

    * Tumor documented to be KRAS WT by local assessment according to institutional standards. If KRAS WT is not previously documented and if archival tissue is not available for pretrial assessment, patient must be willing to undergo a tumor biopsy to confirm eligibility.
    * Confirmed MET-amplification by local assessment.
    * No prior therapy with MET-targeting agents (except a subset of patients having received prior therapy with a MET-targeting TKI).
    * Willingness to undergo a pre- and post-dosing biopsy (maximum of 2 biopsies) from primary or metastatic tumor site(s) considered safely accessible for biopsy
  * NSCLC MET-Amplified Cohort ONLY:

    * Documented NSCLC meeting disease criteria as defined per protocol.
    * Documented MET-amplification.
    * May have received prior therapy with MET-targeting and/or EGFR-targeting agents (antibodies or TKIs).
    * Willingness to undergo a pre-dosing biopsy (mandatory unless a recent tumor biopsy is available), and potentially a biopsy at the End of Cycle 2 (EOC2) (optional), from a primary or metastatic tumor site considered safely accessible for biopsy.
  * NSCLC METex14del Cohort ONLY:

    * Documented NSCLC meeting disease criteria as defined per protocol.
    * Documented METex14del (tumors need not be MET-amplified).
    * May have received prior therapy with MET-targeting and/or EGFR-targeting agents (antibodies or TKIs).
    * Willingness to undergo a pre-dosing biopsy (mandatory unless a recent tumor biopsy is available), and potentially a biopsy at the EOC2 (optional), from a primary or metastatic tumor site considered safely accessible for biopsy.

Exclusion Criteria:

* Any antineoplastic agent for the primary malignancy (standard or investigational) without delayed toxicity within 4 weeks or 5 plasma half-lives, whichever is shortest, prior to C1/D1, except nitrosoureas and mitomycin C within 6 weeks prior to C1/D1.
* Immunosuppressive or systemic hormonal therapy within 2 weeks prior to C1/D1, with exceptions.
* Use of hematopoietic growth factors within 2 weeks prior to C1/D1.
* Active second malignancy or history of another malignancy within the last 3 years, with exceptions.
* Central nervous system (CNS) malignancy including primary malignancies of the CNS and known, untreated CNS or leptomeningeal metastases, or spinal cord compression; patients with any of these not controlled by prior surgery or radiotherapy, or symptoms suggesting CNS involvement for which treatment is required.
* Inadequate recovery from an acute toxicity associated with any prior antineoplastic therapy.
* Major surgical procedure within 4 weeks prior to C1/D1 or inadequate recovery from any prior surgical procedure.
* Active thrombosis, or a history of deep vein thrombosis or pulmonary embolism, within 1 month prior to C1/D1, unless adequately treated and stable.
* Active uncontrolled bleeding or a known bleeding diathesis.
* Significant cardiovascular disease or condition.
* Abnormal hematologic, renal or hepatic function.
* Part 2 ONLY:

  * Radiotherapy against target lesions within 4 weeks prior to C1/D1, unless there is documented progression of the lesion following the radiotherapy.
  * Basket Cohort ONLY:

    * Prior therapy with MET-inhibiting agents (exceptions will be a subset of patients that will be entered to the Basket Cohort after having received prior therapy with a MET-targeting TKI).
    * Prior therapy with antibody to hepatocyte growth factor (HGF).
  * Basket Cohort and NSCLC MET-Amplified Cohort ONLY:

    * Tumor status demonstrating MET-polysomy in the absence of MET-amplification, as specified per protocol. Patients in the NSCLC METex14del Cohort with polysomy are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amita Patnaik, MD, FRCP(C), Principal Investigator — South Texas Accelerated Research Therapeutics, LLC; David Ross Camidge, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (27):
- United States (10):
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute/D -1251, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
- Rigshospitalet, Copenhagen, Denmark
- Queen Mary Hospital, Hong Kong, Hong Kong
- South Korea (6):
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (4):
  - Hospital Universitario Quiron Dexeus, Barcelona, Barcelona/Cataluna
  - Hospital Universitario Vall d'Hebron, Barcelona, Barcelona/Cataluna
  - Hospital Clinic de Barcelona, Barcelona, Barcelona/Cataluna
  - Centro Oncologico MD Anderson, Madrid
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Medical University Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grandal MM, Havrylov S, Poulsen TT, Koefoed K, Dahlman A, Galler GR, Conrotto P, Collins S, Eriksen KW, Kaufman D, Woude GFV, Jacobsen HJ, Horak ID, Kragh M, Lantto J, Bouquin T, Park M, Pedersen MW. Simultaneous Targeting of Two Distinct Epitopes on MET Effectively Inhibits MET- and HGF-Driven Tumor Growth by Multiple Mechanisms. Mol Cancer Ther. 2017 Dec;16(12):2780-2791. doi: 10.1158/1535-7163.MCT-17-0374. Epub 2017 Aug 11. PMID 28802255

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Dose-Escalation; Period 1: 6 mg/kg: Patients received 6 mg/kg Symp015.
  Sym015 was tested in four dose titration cohorts. Patients received increasing doses of 6, 12, 18 and 24 mg/kg every second week (Q2W). A substitute or an additional dose level could potentially be evaluated.
  Dose-escalation followed a standard 3+3 design with escalation dependent upon the occurrence of dose level toxicity.
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
- Part 1: Dose-Escalation; Period 2: 12mg/kg: Patients received 12 mg/kg Symp015.
  Sym015 was tested in four dose titration cohorts. Patients received increasing doses of 6, 12, 18 and 24 mg/kg every second week (Q2W). A substitute or an additional dose level could potentially be evaluated.
  Dose-escalation followed a standard 3+3 design with escalation dependent upon the occurrence of dose level toxicity.
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
- Part 1: Dose-Escalation; Period 3:18mg/kg: Patients received 18 mg/kg Symp015.
  Sym015 was tested in four dose titration cohorts. Patients received increasing doses of 6, 12, 18 and 24 mg/kg every second week (Q2W). A substitute or an additional dose level could potentially be evaluated.
  Dose-escalation followed a standard 3+3 design with escalation dependent upon the occurrence of dose level toxicity.
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
- Part 1: Dose-Escalation; Period 4: 24 mg/kg: Patients received 24 mg/kg Symp015-.
  Sym015 was tested in four dose titration cohorts. Patients received increasing doses of 6, 12, 18 and 24 mg/kg every second week (Q2W). A substitute or an additional dose level could potentially be evaluated.
  Dose-escalation followed a standard 3+3 design with escalation dependent upon the occurrence of dose level toxicity.
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
- Part 2: Dose-Expansion, Basket Cohort: During Part 2, three Cohorts received Sym015 at the recommended phase 2 dose on a every second week dosing schedule:
  Basket Cohort:
  Patients with KRAS proto-oncogene wild-type (KRAS WT) advanced solid tumor malignancies with MET-amplification received Sym015 at the recommended Phase 2 dose. Included in this group was a subset of patients who received prior therapy with a MET-targeting tyrosine kinase inhibitor (TKI).
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
- Part 2: Dose-Expansion, NSCLC MET-Amplified Cohort: During Part 2, three Cohorts received Sym015 at the recommended phase 2 dose on a every second week dosing schedule:
  NSCLC MET-Amplified Cohort:
  Patients with advanced NSCLC with MET-amplification were to receive Sym015 at the RP2D. Patients may have received prior therapy with METtargeting and/or EGFR-targeting agents.
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
- Part 2: Dose-Expansion, NSCLC METEx14Del Cohort: During Part 2, three Cohorts received Sym015 at the recommended phase 2 dose on a every second week dosing schedule:
  NSCLC METex14del Cohort:
  Patients with advanced NSCLC with METex14del were to receive Sym015 at the RP2D. Tumors need not be MET-amplified, and patients may have received prior therapy with MET-targeting and/or EGFR-targeting agents. mutation.
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
Period: Overall Study
Arm/Group | Part 1: Dose-Escalation; Period 1: 6 mg/kg | Part 1: Dose-Escalation; Period 2: 12mg/kg | Part 1: Dose-Escalation; Period 3:18mg/kg | Part 1: Dose-Escalation; Period 4: 24 mg/kg | Part 2: Dose-Expansion, Basket Cohort | Part 2: Dose-Expansion, NSCLC MET-Amplified Cohort | Part 2: Dose-Expansion, NSCLC METEx14Del Cohort
Started | 3 | 3 | 3 | 3 | 25 | 8 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 25 | 8 | 12
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Progressive disease | 2 | 2 | 2 | 3 | 22 | 7 | 8
Not completed — Other reason (unknown) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Transferred to named patient program | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Dose-Escalation, 6 mg/kg; Part 1: Dose-Escalation, 12 mg/kg; Part 1: Dose-Escalation 18 mg/kg; Part 1: Dose-Escalation 24 mg/kg: Sym015 was tested in four dose titration cohorts. A substitute or an additional dose level could potentially be evaluated.
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
- Part 2: Dose-Expansion, Basket Cohort: Patients with KRAS proto-oncogene wild-type (KRAS WT) advanced solid tumor malignancies with MET-amplification received Sym015 at the recommended Phase 2 dose. Included in this group was a subset of patients who received prior therapy with a MET-targeting tyrosine kinase inhibitor (TKI).
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
- Part 2: Dose-Expansion, NSCLC MET-Amplified Cohort: Patients with advanced NSCLC with MET-amplification received Sym015 at the RP2D. Patients may have received prior therapy with METtargeting and/or EGFR-targeting agents.
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
- Part 2: Dose-Expansion, NSCLC METex14del Cohort: Patients with advanced NSCLC with METex14del received Sym015 at the RP2D. Tumors need not be MET-amplified, and patients may have received prior therapy with MET-targeting and/or EGFR-targeting agents.
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
- Total: Total of all reporting groups
Arm/Group | Part 1: Dose-Escalation, 6 mg/kg | Part 1: Dose-Escalation, 12 mg/kg | Part 1: Dose-Escalation 18 mg/kg | Part 1: Dose-Escalation 24 mg/kg | Part 2: Dose-Expansion, Basket Cohort | Part 2: Dose-Expansion, NSCLC MET-Amplified Cohort | Part 2: Dose-Expansion, NSCLC METex14del Cohort | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 25 | 8 | 12 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (14.57) | 62.0 (11.79) | 55.3 (11.24) | 67.3 (7.23) | 56.6 (11.87) | 65.6 (8.91) | 68.5 (9.82) | 61.1 (11.73)
Age, Customized [Count of Participants; unit: Participants]
  18-65 years | 2 | 1 | 2 | 1 | 20 | 2 | 6 | 34
  65 to <75 years | 1 | 2 | 1 | 2 | 4 | 5 | 0 | 15
  75 to <85 years | 0 | 0 | 0 | 0 | 1 | 1 | 6 | 8
  85 years or older | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 7 | 5 | 6 | 25
  Male | 2 | 1 | 1 | 1 | 18 | 3 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 4
  Not Hispanic or Latino | 3 | 3 | 3 | 1 | 24 | 8 | 11 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 14 | 2 | 1 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  White | 2 | 3 | 3 | 2 | 8 | 6 | 11 | 35
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  South Korea | 0 | 0 | 0 | 0 | 12 | 2 | 0 | 14
  United States | 3 | 3 | 3 | 3 | 6 | 3 | 8 | 29
  Taiwan | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Denmark | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Spain | 0 | 0 | 0 | 0 | 6 | 2 | 3 | 11
Body weight [Mean (Standard Deviation); unit: kg] | 82.2 (17.86) | 62.5 (12.03) | 89.0 (18.29) | 69.7 (8.05) | 67.1 (10.73) | 60.3 (11.58) | 72.1 (15.54) | 69.1 (13.86)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg per square meter] — Population: BMI was not evaluable for all participants
  kg per square meter | 28.10 (1.132) | 23.65 (3.978) | 29.84 (7.452) | 25.89 (5.363) | 23.58 (3.776) | 22.15 (4.590) | 25.19 (4.081) | 24.44 (4.405)
ECOG-PS [Count of Participants; unit: Participants] — ECOG-PS=Eastern Cooperative Oncology Group performance status. It describes patient functioning level on a 5 graded scale.
  Grade 0: Fully active, able to carry on all pre-disease performance without restriction Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours Grade 3-5: Ranges from capable of only limited selfcare to dead.
  Participants
    0 | 1 | 2 | 1 | 0 | 4 | 2 | 1 | 11
    1 | 2 | 1 | 2 | 3 | 21 | 6 | 9 | 44
    2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Site of primary tumor [Count of Participants; unit: Participants]
  Breast | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Colon | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 5
  Genitourinary | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 5
  Hepatic (including gallbladder) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Liver | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
  Neck | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Other locally advanced sites | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 5
  Other metastatic sites | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3
  Pancreas | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Respiratory | 0 | 0 | 0 | 0 | 0 | 7 | 12 | 19
  Skin/soft tissue | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Gastrointestinal | 0 | 0 | 0 | 0 | 11 | 0 | 0 | 11
Histopathologic diagnosis [Count of Participants; unit: Participants]
  Adenocarcinoma | 3 | 1 | 1 | 2 | 22 | 7 | 11 | 47
  Missing | 0 | 2 | 2 | 1 | 3 | 1 | 1 | 10
Anatomic based cancer type [Count of Participants; unit: Participants]
  Adenocarcinoma of Parotid Gland | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Adenocarcinoma of Thymus | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  BRCA (breast cancer gene) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  CRC (colorectal cancer) | 2 | 1 | 0 | 0 | 3 | 0 | 0 | 6
  Cholangiocarcinoma | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  GC (gastric cancer) | 0 | 0 | 0 | 0 | 13 | 0 | 0 | 13
  GU (genitourinary cancer) | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 5
  HCC (hepatocellular carcinoma) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  HCC-MIXED | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  HCC-Neuroendocrine | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Lung-Neuroendocrine | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  NSCLC (non-small-cell lung carcinoma) | 0 | 0 | 0 | 0 | 0 | 7 | 11 | 18
  NSCLC- Sq type | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Nasopharyngeal carcinoma | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Pancreatic cancer | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  SCC (squamous cell carcinoma) of skin/soft tissue | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Time since initial diagnosis [Mean (Standard Deviation); unit: years] — Population: Data were not available for all patients in Part 2
  years | 4.7 (2.52) | 2.3 (1.53) | 10.3 (9.29) | 2.0 (2.0) | 2.1 (2.20) | 0 (0) | 0 (0) | 3.5 (4.57)
Previous debulking surgery [Count of Participants; unit: Participants]
  No | 3 | 1 | 2 | 3 | 16 | 7 | 12 | 44
  Yes | 0 | 2 | 1 | 0 | 9 | 1 | 0 | 13
Sites with metastasis [Count of Participants; unit: Participants]
  Abdomen, pelvis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Abdominal cavity, diaphragm, subcutis, para- renal mass, Sub-Hepatic Mass | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Adrenal gland | 0 | 0 | 1 | 0 | 4 | 1 | 4 | 10
  Bone | 1 | 0 | 2 | 2 | 6 | 2 | 7 | 20
  Both ovaries, peritoneum, colon | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Brain | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 5
  Duodenum | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Effusion | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Kidney | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Liver | 2 | 2 | 0 | 2 | 8 | 1 | 2 | 17
  Lungs | 1 | 2 | 2 | 2 | 8 | 7 | 9 | 31
  Lymph nodes | 2 | 3 | 0 | 3 | 20 | 6 | 7 | 41
  Lymph nodes and Lymphangitis Carcinomatoses | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Muscle | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Pelvis, abdominal wall, spleen | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Peritoneal | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Peritoneum, peribiliary | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Pleura | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Pleural based metastases | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Primary gastric cancer | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Rectum | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Skin | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Soft tissue | 0 | 1 | 1 | 1 | 2 | 0 | 3 | 8
  Spleen, pelvis, abdomen, left ovary | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Subpleura | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Thyroid gland | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Number of sites with metastasis [Count of Participants; unit: Participants]
  0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  1 | 1 | 0 | 1 | 0 | 7 | 2 | 1 | 12
  2 | 1 | 0 | 0 | 0 | 8 | 1 | 3 | 13
  3 | 0 | 2 | 1 | 1 | 6 | 3 | 4 | 17
  More than 3 | 1 | 1 | 1 | 2 | 4 | 2 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Occurrence of DLTs During Cycle 1 of Sym015 Administration
Description: The primary objective of Part 1 was to assess the safety and tolerability of Sym015 on a Q2W schedule. This was assessed by evaluating the occurrence of dose-limiting toxicities (DLTs) during Cycle 1 of Sym015 administration. Q2W = every second week.
Time Frame: Cycle 1, the initial 28-day period of Q2W dosing
Population: For evaluation of DLTs, the DLT analysis set was used. This comprised all patients enrolled in Part 1 who had received at least one dose of Sym015, except patients who did not complete Cycle 1 (i.e., the initial 28-day period of Q2W dosing) for reasons other than drug toxicity.
Measure: Number; unit: Number of DLTs
Groups:
- Part 1: Dose-Escalation; Period 1, 6 mg/kg: Patients received 6 mg/kg Sym015.
  Sym015 was tested in four dose titration cohorts. A substitute or an additional dose level could potentially be evaluated.
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
Arm/Group | Part 1: Dose-Escalation; Period 1, 6 mg/kg | Part 1: Dose-Escalation; Period 2: 12mg/kg | Part 1: Dose-Escalation; Period 3:18mg/kg | Part 1: Dose-Escalation; Period 4: 24 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3
Number of DLTs | 0 | 0 | 0 | 0

2. Primary Outcome: Part 2: Documented, Confirmed Objective Response (OR)
Description: The primary objective of Part 2 was to evaluate the antitumor activity of Sym015 when administered at the Q2W RP2D to patients in the different cohorts. Documented OR was defined as partial response [PR] or complete response [CR]) as assessed by CT or MRI using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at any time during trial participation by Investigator assessment. PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; CR = Disappearance of all non-target lesions and normalisation of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  Q2W = every second week. RP2D = recommended phase 2 dose.
Time Frame: 24 months
Population: The Full Analysis Set (FAS) comprised all enrolled patients who had received at least one dose of Sym015.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Basket Cohort: Patients with KRAS proto-oncogene wild-type (KRAS WT) advanced solid tumor malignancies with MET-amplification received Sym015 at the recommended Phase 2 dose. Included in this group was a subset of patients who received prior therapy with a MET-targeting tyrosine kinase inhibitor (TKI).
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
- Part 2: Patients in NSCLC MET-Amplified Cohort: Patients had MET-amplified advanced NSCLC without available therapeutic options. Patients could have received prior therapy with MET-targeting and/or epidermal growth factor receptor (EGFR)-targeting agents.
  NSCL = non-small cell lung cancer. MET = MET proto-oncogene tyrosine kinase, hepatocyte growth factor receptor.
- Part 2: Patients in NSCLC METEx14Del Cohort: Patients had advanced NSCLC with METEx14Del, and without available therapeutic options. Tumors did not need to be MET-amplified, and patients may have received prior therapy with MET-targeting and/or EGFR-targeting agents. NSCLC = non-small cell lung cancer. METEx14Del = MET exon 14 skipping alteration. EGFR = epidermal growth factor receptor.
Arm/Group | Part 2: Basket Cohort | Part 2: Patients in NSCLC MET-Amplified Cohort | Part 2: Patients in NSCLC METEx14Del Cohort
Number analyzed (Participants) | 25 | 8 | 12
Participants | 0 | 2 | 3

3. Secondary Outcome: Part 1: Determine a Q2W RP2D of Sym015.
Description: Determination based on an evaluation of the patient data for DLTs from Part 1. Q2W = every second week. RP2D = recommended phase 2 dose.
Time Frame: 12 Months
Population: It was not possible to determine this endpoint as no DLTs were observed. The RP2D combination was not established and was instead chosen based on other safety findings as well as pharmacokinetic data, as described in the protocol.
Measure: Number; unit: mg/kg
Groups:
- Part 1: Dose-Escalation (4 Arms Combined): Sym015 was tested in four dose titration cohorts (6, 12, 18 and 24 mg/kg) with 3 patients per dose level. A substitute or an additional dose level could potentially be evaluated.
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
Arm/Group | Part 1: Dose-Escalation (4 Arms Combined)
Number analyzed (Participants) | 12
mg/kg | NA — RP2D was not established as no DLTs were observed.

4. Secondary Outcome: Immunogenicity of Sym015: Part 1.
Description: Serum sampling was done to assess the potential for anti-drug antibody (ADA) formation.
Time Frame: Cycle 1: Day (D) 1, Cycle 3, 5, 7: D1 (+-2), End of treatment: At or by D10, Follow-up: 1 month after last dose of study treatment (30+7D)
Population: The Full Analysis Set (FAS) comprised all enrolled patients who had received at least one dose of Sym015.
Measure: Count of Participants; unit: Participants
Groups:
- 6 mg/kg: Cohort of subjects receiving a dose of 6 mg/kg of Sym015 administered by intravenous infusion Q2W. Q2W = every second week.
- 12 mg/kg: Cohort of subjects receiving a dose of 12 mg/kg of Sym015 administered by intravenous infusion Q2W. Q2W = every second week.
- 18 mg/kg: Cohort of subjects receiving a dose of 18 mg/kg of Sym015 administered by intravenous infusion Q2W. Q2W = every second week.
- 24 mg/kg: Cohort of subjects receiving a dose of 24 mg/kg of Sym015 administered by intravenous infusion Q2W. Q2W = every second week.
Arm/Group | 6 mg/kg | 12 mg/kg | 18 mg/kg | 24 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants
  Cycle 1 - day 1: Not done | 0 | 0 | 0 | 0
  Cycle 1 - day 1: Negative | 3 | 3 | 3 | 3
  Cycle 1 - day 1: Patient withdrawn | 0 | 0 | 0 | 0
  Cycle 3 - day 1: Not done | 0 | 0 | 0 | 0
  Cycle 3 - day 1: Negative | 1 | 0 | 2 | 0
  Cycle 3 - day 1: Patient withdrawn | 2 | 3 | 1 | 3
  End of treatment: Not done | 0 | 0 | 0 | 1
  End of treatment: Negative | 3 | 2 | 1 | 2
  End of treatment: Patient withdrawn | 0 | 1 | 2 | 0
  1-month follow-up: Not done | 0 | 1 | 0 | 0
  1-month follow-up: Negative | 2 | 1 | 0 | 2
  1-month follow-up: Patient withdrawn | 1 | 1 | 3 | 1

5. Secondary Outcome: Immunogenicity of Sym015: Part 2.
Description: Serum sampling was done to assess the potential for anti-drug antibody (ADA) formation.
Time Frame: Cycle 1: Day (D) 1, Cycle 2, 3, 5, 7: D1 (+-2), End of treatment: At or by D10, Follow-up: 1 month after last dose of study treatment (30+7D)
Population: The Full Analysis Set (FAS) comprised all enrolled patients who had received at least one dose of Sym015.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Basket Cohort | Part 2: Patients in NSCLC MET-Amplified Cohort | Part 2: Patients in NSCLC METEx14Del Cohort
Number analyzed (Participants) | 25 | 8 | 12
Participants
  Cycle 1 - day 1: Not done | 0 | 0 | 0
  Cycle 1 - day 1: Negative | 25 | 8 | 12
  Cycle 1 - day 1: Positive | 0 | 0 | 0
  Cycle 1 - day 1: Patient withdrawn | 0 | 0 | 0
  Cycle 2 - day 1: Not done | 1 | 0 | 0
  Cycle 2 - day 1: Negative | 21 | 8 | 11
  Cycle 2 - day 1: Positive | 0 | 0 | 0
  Cycle 2 - day 1: Patient withdrawn | 3 | 0 | 1
  Cycle 3 - day 1: Not done | 1 | 1 | 0
  Cycle 3 - day 1: Negative | 8 | 7 | 8
  Cycle 3 - day 1: Positive | 0 | 0 | 0
  Cycle 3 - day 1: Patient withdrawn | 16 | 0 | 4
  Cycle 5 - day 1: Not done | 0 | 0 | 1
  Cycle 5 - day 1: Negative | 6 | 6 | 5
  Cycle 5 - day 1: Positive | 0 | 0 | 0
  Cycle 5 - day 1: Patient withdrawn | 19 | 2 | 6
  Cycle 7 - day 1: Not done | 0 | 1 | 0
  Cycle 7 - day 1: Negative | 2 | 2 | 5
  Cycle 7 - day 1: Positive | 0 | 0 | 0
  Cycle 7 - day 1: Patient withdrawn | 23 | 5 | 7
  End of treatment: Not done | 5 | 0 | 0
  End of treatment: Negative | 15 | 7 | 9
  End of treatment: Positive | 1 | 0 | 0
  End of treatment: Patient withdrawn | 4 | 1 | 3
  1-month follow up: Not done | 0 | 1 | 1
  1-month follow up: Negative | 10 | 3 | 5
  1-month follow up: Positive | 1 | 0 | 0
  1-month follow up: Patient withdrawn | 14 | 4 | 6

6. Secondary Outcome: Part 1: Area Under the Concentration-time Curve in a Dosing Interval (AUC) Following 1st Dose
Description: Estimated using non-compartmental methods and actual time points following the first dose of Sym015.
Time Frame: From time zero to 48 hours after dosing. Samples taken pre-dosing and at 1, 2, 4, 8, 24 and 48 hours after end of infusion.
Measure: Median (Full Range); unit: h*μg/mL
Arm/Group | 6 mg/kg | 12 mg/kg | 18 mg/kg | 24 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3
h*μg/mL | 17900 [17100 to 24500] | 35700 [31600 to 42900] | 82500 [75200 to 86200] | 76800 [55200 to 86400]

7. Secondary Outcome: Part 2: Area Under the Concentration-time Curve in a Dosing Interval (AUC)
Description: Estimated using non-compartmental methods and actual time points following the first dose of Sym015 for the whole basket cohort.
Time Frame: as for outcome 6
Measure: Median (Full Range); unit: h*ug/mL
Groups:
- Part 2 (Dose Expansion): Basket Cohort: Patients with KRAS proto-oncogene wild-type (KRAS WT) advanced solid tumor malignancies with MET-amplification received Sym015 at the recommended Phase 2 dose: 18 mg/kg loading dose followed by 12 mg/kg Q2W maintenance dose.
  Included in this group was a subset of patients who received prior therapy with a MET-targeting tyrosine kinase inhibitor (TKI).
- Part 2 (Dose Expansion): Patients in NSCLC MET-Amplified Cohort: Patients had MET-amplified advanced NSCLC without available therapeutic options. Patients could have received prior therapy with MET-targeting and/or epidermal growth factor receptor (EGFR)-targeting agents.
  Sym015 was administered at the recommended Phase 2 dose: 18 mg/kg loading dose followed by 12 mg/kg Q2W maintenance dose.
  NSCL = non-small cell lung cancer. MET = MET proto-oncogene tyrosine kinase, hepatocyte growth factor receptor.
- Part 2 (Dose Expansion): Patients in NSCLC METEx14Del Cohort: Patients had advanced NSCLC with METEx14Del, and without available therapeutic options. Tumors did not need to be MET-amplified, and patients may have received prior therapy with MET-targeting and/or EGFR-targeting agents.
  Sym015 was administered at the recommended Phase 2 dose: 18 mg/kg loading dose followed by 12 mg/kg Q2W maintenance dose.
  NSCLC = non-small cell lung cancer. METEx14Del = MET exon 14 skipping alteration. EGFR = epidermal growth factor receptor.
Arm/Group | Part 2 (Dose Expansion): Basket Cohort | Part 2 (Dose Expansion): Patients in NSCLC MET-Amplified Cohort | Part 2 (Dose Expansion): Patients in NSCLC METEx14Del Cohort
Number analyzed (Participants) | 25 | 8 | 12
h*ug/mL | 34000 [17300 to 51800] | 37200 [22000 to 55000] | 38700 [11300 to 54000]

8. Secondary Outcome: Part 1: Cmax
Description: Maximum serum concentration was derived from observed data.
Time Frame: as for outcome 6
Measure: Median (Full Range); unit: ug/mL
Arm/Group | 6 mg/kg | 12 mg/kg | 18 mg/kg | 24 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3
ug/mL | 146 [141 to 151] | 286 [275 to 323] | 563 [419 to 711] | 561 [379 to 726]

9. Secondary Outcome: Part 2: Cmax
Description: Maximum serum concentration was derived from observed data following the first dose of Sym015 for the full basket cohort.
Time Frame: as for outcome 6
Measure: Median (Full Range); unit: ug/mL
Groups:
- Part 2 (Dose-Expansion): Basket Cohort: Patients with KRAS proto-oncogene wild-type (KRAS WT) advanced solid tumor malignancies with MET-amplification received Sym015 at the recommended Phase 2 dose: 18 mg/kg loading dose followed by 12 mg/kg Q2W maintenance dose.. Included in this group was a subset of patients who received prior therapy with a MET-targeting tyrosine kinase inhibitor (TKI).
- Part 2 (Dose-Expansion): Patients in NSCLC MET-Amplified Cohort: Patients had MET-amplified advanced NSCLC without available therapeutic options. Patients could have received prior therapy with MET-targeting and/or epidermal growth factor receptor (EGFR)-targeting agents.
  Sym015 was administered at the recommended Phase 2 dose: 18 mg/kg loading dose followed by 12 mg/kg Q2W maintenance dose.
  NSCL = non-small cell lung cancer. MET = MET proto-oncogene tyrosine kinase, hepatocyte growth factor receptor.
- Part 2 (Dose-Expansion): Patients in NSCLC METEx14Del Cohort: Patients had advanced NSCLC with METEx14Del, and without available therapeutic options. Tumors did not need to be MET-amplified, and patients may have received prior therapy with MET-targeting and/or EGFR-targeting agents.
  Sym015 was administered at the recommended Phase 2 dose: 18 mg/kg loading dose followed by 12 mg/kg Q2W maintenance dose.
  NSCLC = non-small cell lung cancer. METEx14Del = MET exon 14 skipping alteration. EGFR = epidermal growth factor receptor.
Arm/Group | Part 2 (Dose-Expansion): Basket Cohort | Part 2 (Dose-Expansion): Patients in NSCLC MET-Amplified Cohort | Part 2 (Dose-Expansion): Patients in NSCLC METEx14Del Cohort
Number analyzed (Participants) | 25 | 8 | 12
ug/mL | 420 [310 to 700] | 520 [320 to 610] | 510 [330 to 1180]

10. Secondary Outcome: Part 1: Time to Reach Maximum Concentration (Tmax)
Description: Time to reach maximum concentration (Tmax) was derived from observed data.
Time Frame: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | 6 mg/kg | 12 mg/kg | 18 mg/kg | 24 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3
hours | 2.1 [2 to 5] | 1.1 [1 to 2] | 3.5 [3 to 4] | 3.0 [3 to 9]

11. Secondary Outcome: Part 2: Time to Reach Maximum Concentration (Tmax)
Description: Time to reach maximum concentration (Tmax) was derived from observed data following the first dose of Sym015 for the full basket cohort.
Time Frame: as for outcome 6
Measure: Median (Full Range); unit: hours
Groups:
- Part 2 (Dose-Expansion): Basket Cohort: Patients with KRAS proto-oncogene wild-type (KRAS WT) advanced solid tumor malignancies with MET-amplification received Sym015 at the recommended Phase 2 dose: 18 mg/kg loading dose followed by 12 mg/kg Q2W maintenance dose.. Included in this group was a subset of patients who received prior therapy with a MET-targeting tyrosine kinase inhibitor (TKI).
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
Arm/Group | Part 2 (Dose-Expansion): Basket Cohort | Part 2 (Dose-Expansion): Patients in NSCLC MET-Amplified Cohort | Part 2 (Dose-Expansion): Patients in NSCLC METEx14Del Cohort
Number analyzed (Participants) | 25 | 8 | 12
hours | 2.5 [1 to 44] | 3.7 [2 to 8] | 2.8 [2 to 7]

12. Secondary Outcome: Part 1: Trough Concentration (Ctrough)
Description: Ctrough was derived from observed data.
Time Frame: as for outcome 6
Measure: Median (Full Range); unit: μg/mL
Arm/Group | 6 mg/kg | 12 mg/kg | 18 mg/kg | 24 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3
μg/mL | 23.1 [19.2 to 31.5] | 61.3 [56.1 to 65] | 130 [127 to 187] | 92.4 [91.3 to 151]

13. Secondary Outcome: Part 2: Trough Concentration (Ctrough)
Description: Ctrough was derived from observed data following the first dose of Sym015 for the whole basket cohort.
Time Frame: as for outcome 6
Measure: Median (Full Range); unit: μg/mL
Arm/Group | Part 2 (Dose-Expansion): Basket Cohort | Part 2 (Dose-Expansion): Patients in NSCLC MET-Amplified Cohort | Part 2 (Dose-Expansion): Patients in NSCLC METEx14Del Cohort
Number analyzed (Participants) | 24 | 8 | 11
μg/mL | 84.1 [24 to 429] | 90.1 [51 to 183] | 101.7 [66 to 250]

14. Secondary Outcome: Part 1: Elimination Half-life (T½)
Description: Estimated using non-compartmental methods and actual time points.
Time Frame: as for outcome 6
Population: Numbers reflects evaluable participants. Evaluable participants = T½ is only reported if at least three data points were available in the terminal phase, R2 in 0.85 or above and the time span between the first and the last data point for z covers at least 1.5 half-lives. Reference: V-QUAL-107812
Measure: Median (Full Range); unit: hours
Arm/Group | 6 mg/kg | 12 mg/kg | 18 mg/kg | 24 mg/kg
Number analyzed (Participants) | 3 | 1 | 1 | 1
hours | 179 [116 to 179] | 137 [137 to 137] | 193 [193 to 193] | 170 [170 to 170]

15. Secondary Outcome: Part 2: Elimination Half-life (T½)
Description: as for outcome 7
Time Frame: as for outcome 6
Measure: Median (Full Range); unit: hours
Groups:
- Part 2 (Dose-Expansion): Basket Cohort: Patients with KRAS proto-oncogene wild-type (KRAS WT) advanced solid tumor malignancies with MET-amplification received Sym015 at the recommended Phase 2 dose: 18 mg/kg loading dose followed by 12 mg/kg Q2W maintenance dose. Included in this group was a subset of patients who received prior therapy with a MET-targeting tyrosine kinase inhibitor (TKI).
Arm/Group | Part 2 (Dose-Expansion): Basket Cohort | Part 2 (Dose-Expansion): Patients in NSCLC MET-Amplified Cohort | Part 2 (Dose-Expansion): Patients in NSCLC METEx14Del Cohort
Number analyzed (Participants) | 13 | 6 | 7
hours | 150 [87 to 217] | 191 [103 to 208] | 171 [116 to 204]

16. Secondary Outcome: Part 1: Clearance (CL)
Description: Estimated using non-compartmental methods and actual time points.
Time Frame: as for outcome 6
Population: Samples were determined for subjects in the 6 and 12 mg/kg cohorts. No samples from subjects in the 18 and 24 mg/kg cohorts were available for analysis.
Measure: Median (Full Range); unit: mL/h
Arm/Group | 6 mg/kg | 12 mg/kg | 18 mg/kg | 24 mg/kg
Number analyzed (Participants) | 1 | 1 | 0 | 0
mL/h | 0.3 [0.3 to 0.3] | 0.2 [0.2 to 0.2] |  |

17. Secondary Outcome: Part 2: Clearance (CL)
Description: as for outcome 7
Time Frame: as for outcome 6
Measure: Median (Full Range); unit: mL/h/kg
Groups:
- Part 2 (Dose-Expansion): Basket Cohort: Patients with KRAS proto-oncogene wild-type (KRAS WT) advanced solid tumor malignancies with MET-amplification received Sym015 at the recommended Phase 2 dose: 18 mg/kg loading dose followed by 12 mg/kg Q2W maintenance dose. Included in this group was a subset of patients who received prior therapy with a MET-targeting tyrosine kinase inhibitor (TKI).
  Sym015: Sym015 is a mixture of two monoclonal antibodies which specifically bind to non-overlapping epitopes in the extracellular domain of MET.
Arm/Group | Part 2 (Dose-Expansion): Basket Cohort | Part 2 (Dose-Expansion): Patients in NSCLC MET-Amplified Cohort | Part 2 (Dose-Expansion): Patients in NSCLC METEx14Del Cohort
Number analyzed (Participants) | 7 | 1 | 2
mL/h/kg | 0.4 [0.2 to 0.5] | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.2]

18. Secondary Outcome: Part 2: Additional Preliminary Evaluation of the Antitumor Activity of Sym015 When Administered at the Q2W RP2D in a Subset of Patients. Assessed by OR.
Description: This applies to the subset of patients in the Basket Cohort who received prior therapy with a MET-targeting TKI. Documented OR (defined as PR or CR), assessed by RECIST v1.1 at any time during trial participation by Investigator assessment.
  Objective Response (OR) is presented. Documented OR was defined as partial response [PR] or complete response [CR]) as assessed by CT or MRI using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at any time during trial participation by Investigator assessment.
  PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; CR = Disappearance of all non-target lesions and normalisation of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Prior MET-targeting TKI Therapy (Basket Cohort): Patients in Basket Cohort, with prior MET-targeting TKI therapy. MET = MET proto-oncogene tyrosine kinase, hepatocyte growth factor receptor. TKI = tyrosine kinase inhibitor.
- Patients Without Prior MET-targeting TKI Therapy (Basket Cohort): Patients in Basket Cohort, without prior MET-targeting TKI therapy. MET = MET proto-oncogene tyrosine kinase, hepatocyte growth factor receptor. TKI = tyrosine kinase inhibitor.
Arm/Group | Patients With Prior MET-targeting TKI Therapy (Basket Cohort) | Patients Without Prior MET-targeting TKI Therapy (Basket Cohort)
Number analyzed (Participants) | 5 | 20
Participants | 0 | 0

19. Secondary Outcome: Part 2: Additional Preliminary Evaluation of the Antitumor Activity of Sym015 When Administered at the Q2W RP2D in a Subset of Patients. Assessed by DCR.
Description: This applies to the subset of patients in the Basket Cohort who received prior therapy with a MET-targeting TKI. Documented OR (defined as PR or CR), assessed by RECIST v1.1 at any time during trial participation by Investigator assessment.
  Disease control rate (DCR) is presented. The DCR was defined as the percentage of patients who had BOR of confirmed CR or confirmed PR or SD (including unconfirmed CR/PR, provided 6 weeks minimum criteria for SD duration was met).
  BOR = Best Overall Response. CR = Complete Response. PR = Partial Response. SD = Stable Disease.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Prior MET-targeting TKI Therapy (Basket Cohort) | Patients Without Prior MET-targeting TKI Therapy (Basket Cohort)
Number analyzed (Participants) | 5 | 20
Participants | 2 | 8

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Part 1: Dose-Escalation; Period 1: 6 mg/kg | Part 1: Dose-Escalation; Period 2: 12mg/kg | Part 1: Dose-Escalation; Period 3:18mg/kg | Part 1: Dose-Escalation; Period 4: 24 mg/kg | Part 2: Dose-Expansion, Basket Cohort | Part 2: Dose-Expansion, NSCLC MET-Amplified Cohort | Part 2: Dose-Expansion, NSCLC METEx14Del Cohort
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/25 | 0/8 | 3/12
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/3 | 1/3 | 8/25 | 4/8 | 6/12
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 3/3 | 3/3 | 23/25 | 8/8 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Dose-Escalation; Period 1: 6 mg/kg (N=3) | Part 1: Dose-Escalation; Period 2: 12mg/kg (N=3) | Part 1: Dose-Escalation; Period 3:18mg/kg (N=3) | Part 1: Dose-Escalation; Period 4: 24 mg/kg (N=3) | Part 2: Dose-Expansion, Basket Cohort (N=25) | Part 2: Dose-Expansion, NSCLC MET-Amplified Cohort (N=8) | Part 2: Dose-Expansion, NSCLC METEx14Del Cohort (N=12)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Dose-Escalation; Period 1: 6 mg/kg (N=3) | Part 1: Dose-Escalation; Period 2: 12mg/kg (N=3) | Part 1: Dose-Escalation; Period 3:18mg/kg (N=3) | Part 1: Dose-Escalation; Period 4: 24 mg/kg (N=3) | Part 2: Dose-Expansion, Basket Cohort (N=25) | Part 2: Dose-Expansion, NSCLC MET-Amplified Cohort (N=8) | Part 2: Dose-Expansion, NSCLC METEx14Del Cohort (N=12)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Presbyesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema peripheral (General disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (6) | 7 (11)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 6 (7) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 2 (2) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Early satiety (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 0 (0) | 3 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 1 (1) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear hemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT02648724/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT02648724/SAP_001.pdf